CLINICAL TRIAL: NCT05484492
Title: Ridge Preservation Comparing the Clinical and Histologic Healing of Two Different Putty Bone Grafts
Brief Title: Alveolar Ridge Preservation With Putty Allograft vs. Putty Alloplast Graft
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Louisville (Other)
Collaborators: BioHorizons, Inc. (Industry)
Responsible Party: Principal Investigator, Himabindu Dukka, Director, Graduate Periodontics, University of Louisville
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 22.0560
Record Dates: First submitted 2022-07-06; First posted 2022-08-02 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-03

CONDITIONS: Alveolar Bone Resorption
Keywords: Alveolar ridge preservation; Socket preservation
MeSH Terms: interventions — Bioglass

STUDY DESIGN:
Intervention Model Description: Thirty patients will be treated using the principles of guided bone regeneration utilizing a full thickness flap for ridge preservation. Fifteen test patients will receive an intrasocket demineralized and mineralized combination putty allograft with a regenerative tissue matrix membrane. The positive control group of fifteen patients will receive an intrasocket synthetic resorbable calcium phosphosilicate putty alloplast graft covered with a regenerative tissue matrix membrane. Approximately four months post-surgery, a trephine core will be taken from the grafted site immediately prior to implant placement and submitted for histologic processing.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The study involves an investigator (surgeon) and an examiner. The examiner measures the clinical parameters before and after surgery and is blinded to the surgical procedure and type of graft the patient receives.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- demineralized and mineralized combination putty bone allograft (Experimental): Fifteen test patients will receive an intrasocket demineralized and mineralized combination putty allograft (MinerOss Putty, BioHorizons) with a regenerative tissue matrix membrane (AlloDerm GBR, BioHorizons) following tooth extraction.
  Interventions: Biological: demineralized and mineralized combination putty bone allograft
- calcium phosphosilicate putty alloplast graft (Active Comparator): The positive control group of fifteen patients will receive an intrasocket synthetic resorbable calcium phosphosilicate putty alloplast graft (NovaBone, Osteogenics) covered with a regenerative tissue matrix membrane (AlloDerm GBR, BioHorizons) following tooth extraction.
  Interventions: Biological: calcium phosphosilicate putty alloplast graft

INTERVENTIONS:
Biological: demineralized and mineralized combination putty bone allograft — Subjects in this group will receive an intrasocket demineralized and mineralized combination putty bone allograft following tooth extraction
  Other Names: MinerOss Putty, BioHorizons
  Arms: demineralized and mineralized combination putty bone allograft
Biological: calcium phosphosilicate putty alloplast graft — Subjects in this group will receive an intrasocket synthetic resorbable calcium phosphosilicate putty alloplast graft following tooth extraction
  Other Names: NovaBone, Osteogenics
  Arms: calcium phosphosilicate putty alloplast graft

SUMMARY:
The primary aims of this study are to compare, after 4 months, the clinical and histologic results of a combination demineralized/mineralized putty allograft vs. synthetic calcium phosphosilicate (CPS) putty alloplast graft utilization in socket preservation procedures. A regenerative tissue matrix membrane will be used to cover each graft lying below the flap.

DETAILED DESCRIPTION:
Study design Thirty patients will be treated using the principles of guided bone regeneration utilizing a full thickness flap for ridge preservation. Fifteen test patients will receive an intrasocket demineralized and mineralized combination putty allograft with a regenerative tissue matrix membrane. The positive control group of fifteen patients will receive an intrasocket synthetic resorbable calcium phosphosilicate putty alloplast graft covered with a regenerative tissue matrix membrane. Approximately, four months post-surgery, a trephine core will be taken from the grafted site immediately prior to implant placement and submitted for histologic processing.

Presurgical Management

Each patient will receive a diagnostic work-up including standardized radiographs (periapical), cone beam computed tomography (CBCT) scan, study casts, clinical photographs, and a clinical examination to record attachment level, probing depth, recession, and mobility of teeth adjacent to the extracted sites. Customized acrylic occlusal stents will be fabricated on the study casts to serve as fixed reference guides for the measurements. Presurgical preparation will include detailed oral hygiene instructions. Baseline data will be collected just before the surgical phase of the treatment. Baseline data will include:

Clinical Measurements

Baseline and 4-month data will include the following:

For the extraction site or adjacent teeth when necessary:

1. Plaque index
2. Gingival index
3. Gingival margin levels: Measured from cemento-enamel junction (CEJ) to the gingival margin.
4. Keratinized tissue: Measured from the gingival margin to the mucogingival junction.
5. Clinical attachment level: Measured from CEJ to the bottom of the clinical periodontal pocket.
6. Clinical tooth mobility: Measured by using the modified Miller's Index.
7. Ridge dimensions: Post-extraction and 4 month healing stent and caliper measurements.
8. Soft tissue thickness.
9. Radiographic examination including CBCT
10. Clinical photographs.

Histologic Measurements

For preservation sites:

1. Trephine core specimens will be evaluated to determine percent vital bone, non-vital bone, and trabecular space. Step serial sections will be taken from each longitudinally sectioned core. The sections will be stained with hematoxylin and eosin. Ten slides per patients will be prepared with at least 4 sections per slide. For each patient, 6 of 10 slides will be assessed. The mean percentage of vital and nonvital bone, and trabecular space will be determined for each patient by using an American Optical microscope at 150X with 10 X 10 ocular grid.

Potential Risks

There are known physical risks linked with tooth extraction with the placement of the bone graft materials (human) in the jaw as well as risks linked with surgical implant placement. The potential risks are the same as the risks of any minor surgery in the mouth. These risks include:

* Infection of treated area (usually mild, rare less than 1%)
* Mild bruising and/or bleeding (less likely 1-39%)
* Mild swelling (more than 40%)
* Transient but occasional paresthesia or numbness of lips, tongue, chin or gum (usually mild, rare less than 1%)
* Loss of the bone graft (mild to moderate, rare less than 1%)

There may also be additional risks that are currently unforeseeable.

Adverse Events Definitions An "adverse event" refers to any adverse experience occurring during the clinical study period, whether associated or not associated with the study test articles or procedures. A "serious adverse event" means any experiences that suggest significant hazard, contraindication, side effect, or precaution. With respect to human clinical experience, a serious adverse event includes any experience that is fatal or life threatening, causes a persistent or permanent disability, requires initial or prolonged hospitalization, requires medical or surgical intervention to prevent permanent impairment or damage, or is a congenital anomaly.

An "unanticipated adverse event" is one that is not identified in nature, severity, or frequency.

Procedure Adverse events will be collected by observing and interviewing the subject during the study. Subjects who experience any significant problems during the study are to call and discuss them with investigator. Any suspected adverse event or allergic response is to be thoroughly examined by investigator. All adverse events are to be reported. All subjects experiencing adverse events will be followed by the investigator until there is a return to the subject's baseline condition or a clinically satisfactory resolution is achieved. Adverse events that are serious or unanticipated are to be reported immediately by phone to the study director and promptly reported to the institutional review board (IRB), which will include the event date, description of the adverse event, study treatment involved, and outcome of event. Examples of expected, but rarely occurring adverse events related to grafting treatment include clinical observation of infection, flap necrosis, severe inflammation, and severe pain.

Measurement techniques All probing measurements will be taken using the University of North Carolina probe. A masked, calibrated examiner will perform the initial examination and the measurements at the time of initial surgery using a customized stent. The mentor will check these measurements. Differences of more than 1.0 mm between examiners will be remeasured by the blinded examiner. Measurements will again be repeated at the 4-month examination using the same techniques.

Statistical Analysis Means and standard deviations will be calculated for all parameters. A paired t-test will be used to evaluate the statistical significance of the differences between initial and final data. An unpaired t-test will be used to evaluate statistical differences between the test and control groups. The sample size of 15 per group gives 83% statistical power to detect a difference of 1 mm between groups. Power calculations were based on data from previous studies.

Research materials, records and privacy: The de-identified data collected will be entered in an excel spreadsheet, which will be password protected. The data will be stored in an encrypted computer, which is also password protected. No one will have access to this data other than the individual collecting it and the PI. No personal identifying information will be collected or needed for the study analytical purposes.

Significance The results of this study will allow comparison of a combination putty allograft versus demineralized putty allograft covered by a regenerative tissue matrix membrane for ridge preservation in terms of the effect on vertical and horizontal dimensions, suitability of the site to receive an implant, and histologic bone quality.

The Plaque Index

The modified O'Leary plaque index (plaque free sites) will be used to obtain dichotomous plaque scores at 6 sites per tooth.

The Gingival Index

The Gingival Index (Lobene et al. 1986) will be measured. Scores will be as follows:

0- Absence of inflammation

1. Mild inflammation; slight change in color, little change in texture of any portion of but not the entire marginal or papillary gingival unit.
2. Mild inflammation; criteria as above but involving the entire marginal or papillary gingival unit.
3. Moderate inflammation; glazing, redness, edema, and/or hypertrophy of the marginal or papillary gingival unit.
4. Severe inflammation; marked redness, edema and/or hypertrophy of the marginal or papillary gingival unit, spontaneous bleeding, congestion, or ulceration.

Each gingival unit (buccal, lingual, mesiobuccal, distobuccal, mesiolingual, and distolingual) of the individual tooth will be given a score from 0-4, called the gingival index for the area. The scores from the 6 areas of the tooth are added and divided by 6 to give the gingival index for the tooth.

Standardized Radiographic technique

An occlusal stent is used to provide a stable foundation for the radiograph holder. The stent is placed on a cast and the Rinn radiograph holder is positioned to allow as near as possible paralleling technique. Radiographs will be taken at baseline and again at 4 months.

Arithmetic determinations:

Change in horizontal ridge dimension: Pre-op width - post-op width

Change in vertical ridge dimension: Pre-op stent distance - Post-op stent distance

Tooth mobility

Miller proposed the following tooth mobility index:

0 - Mobility of the crown is within normal physiologic limits.

1. - Mobility of the crown up to 0.5 mm in one direction. Does not exceed 1.0 mm in both directions.
2. - Mobility of the crown from 0.5 to 1 mm in one direction. Does not exceed 2.0 mm in both directions.
3. - Mobility of the crown exceeding 1 mm in one direction and/or vertical depressibility. Greater than 2.0 mm in both directions and/or vertical depressibility.

The index that will be used in the study is a modification of Miller's index (Laster et al., 1975) where half scores are used. Thus, scores of 0, 0.5, 1, 1.5, 2, 2.5, and 3 will be utilized.

Stent fabrication

Rigid stents will be made of 3 mm thick acrylic plates in order to obtain reproducible measurements. The acrylic will be pressed over a model cast and cured using a curing light so that the edge extends just apical to the prominence of the teeth. Holes will be cut into the splint with a high-speed handpiece in order to allow probing in the needed areas of edentulous ridge in order to produce reproducible probing spots and directions of probe insertions. The holes will be made on the buccal and lingual aspects of the splint for horizontal readings and on the top aspect for vertical readings.

Examiner calibration: Probing and caliper measurements.

The data will be compared from indices or measurements taken by the examiner on three different patients at two different times within a 60-minute period to measure the intra-examiner accuracy and reproducibility.

1. A minimum of three subjects are to be recruited to participate in the calibration. The subjects should exhibit a range of the criteria being assessed in the index or measurements being performed (i.e., subjects with moderate to severe periodontal disease).
2. The examiner will score 3 teeth per subject within the same quadrant.
3. The examiner will measure each subject, calling out the measurements, site by site, while the assistant records.
4. Duplicate measurements of the subjects will be taken within 60 minutes following the initial measurements. The assistant will record the second set of data.
5. The examiner will not compare the two sets of data at any time during the calibration. The examiner will not discuss their measurements with the assistant or the subject during the calibration.
6. The assistant recording the data will be responsible for handling the data sheets. The examiner will have no access to any of the data sheets during the course of the calibration.

8. The data sets will be analyzed for percent agreement. Acceptable percent agreement will reflect the limits set for the different parameters measured.

9. Acceptable percent agreement will be: 90% within ±1mm for probing depth, recession and attachment level and 70% within 0 mm.

ELIGIBILITY:
Inclusion Criteria:

1. Have one non-molar tooth requiring extraction that will be replaced by a dental implant.

   The site must be bordered by at least one tooth.
2. Healthy male or female who is at least 18 years old.
3. Patients must sign an informed consent approved by the University of Louisville Human Studies Committee.

Exclusion Criteria:

1. Patients with debilitating systemic diseases, or diseases that have a clinically significant effect on the periodontium.
2. Presence or history of osteonecrosis of jaws.
3. Patients who are currently taking IV bisphosphonates or who had IV treatment with bisphosphonates irrespective of duration.
4. Patients who have been treated with oral bisphosphonates for more than three years.
5. Patients with an allergy to any material or medication used in the study.
6. Patients who need prophylactic antibiotics
7. Previous head and neck radiation therapy.
8. Chemotherapy in the previous 12 months.
9. Patients on long term NSAID or steroid therapy.
10. Pregnant patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-10-06 (Actual); Primary Completion 2025-10-07 (Actual); Study Completion 2025-10-30 (Actual)

PRIMARY OUTCOMES:
Alveolar ridge width | 4 months
  Alveolar ridge width (measured in mm) after 4 months of healing
Alveolar ridge height | 4 months
  Alveolar ridge height (measured in mm) after 4 months of healing
Buccal soft tissue thickness | 4 months
  Buccal soft tissue thickness at crest of alveolar ridge (measured in mm)

SECONDARY OUTCOMES:
Percentage of vital bone present | 4 months
  Histologic measurement of the percentage of vital bone cells taken from core biopsy of grafted site at 4 months post-op

CONTACTS AND LOCATIONS:
Overall Officials: Bindu Dukka, BDS,MSD,MPH, Principal Investigator — Director, Graduate Periodontics, University of Louisville
Locations (1):
- University of Louisville, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Araujo MG, Lindhe J. Dimensional ridge alterations following tooth extraction. An experimental study in the dog. J Clin Periodontol. 2005 Feb;32(2):212-8. doi: 10.1111/j.1600-051X.2005.00642.x. PMID 15691354
- [Background] Araujo MG, da Silva JCC, de Mendonca AF, Lindhe J. Ridge alterations following grafting of fresh extraction sockets in man. A randomized clinical trial. Clin Oral Implants Res. 2015 Apr;26(4):407-412. doi: 10.1111/clr.12366. Epub 2014 Mar 12. PMID 24621203
- [Background] Barone A, Ricci M, Tonelli P, Santini S, Covani U. Tissue changes of extraction sockets in humans: a comparison of spontaneous healing vs. ridge preservation with secondary soft tissue healing. Clin Oral Implants Res. 2013 Nov;24(11):1231-7. doi: 10.1111/j.1600-0501.2012.02535.x. Epub 2012 Jul 12. PMID 22784417
- [Background] Jung RE, Philipp A, Annen BM, Signorelli L, Thoma DS, Hammerle CH, Attin T, Schmidlin P. Radiographic evaluation of different techniques for ridge preservation after tooth extraction: a randomized controlled clinical trial. J Clin Periodontol. 2013 Jan;40(1):90-8. doi: 10.1111/jcpe.12027. Epub 2012 Nov 19. PMID 23163915
- [Background] Laster L, Laudenbach KW, Stoller NH. An evaluation of clinical tooth mobility measurements. J Periodontol. 1975 Oct;46(10):603-7. doi: 10.1902/jop.1975.46.10.603. PMID 1058939
- [Background] Leblebicioglu B, Salas M, Ort Y, Johnson A, Yildiz VO, Kim DG, Agarwal S, Tatakis DN. Determinants of alveolar ridge preservation differ by anatomic location. J Clin Periodontol. 2013 Apr;40(4):387-95. doi: 10.1111/jcpe.12065. Epub 2013 Feb 21. PMID 23432761
- [Background] Llanos AH, Sapata VM, Jung RE, Hammerle CH, Thoma DS, Cesar Neto JB, Pannuti CM, Romito GA. Comparison between two bone substitutes for alveolar ridge preservation after tooth extraction: Cone-beam computed tomography results of a non-inferiority randomized controlled trial. J Clin Periodontol. 2019 Mar;46(3):373-381. doi: 10.1111/jcpe.13079. Epub 2019 Mar 3. PMID 30710389
- [Background] O'Leary TJ, Drake RB, Naylor JE. The plaque control record. J Periodontol. 1972 Jan;43(1):38. doi: 10.1902/jop.1972.43.1.38. No abstract available. PMID 4500182
- [Background] Lobene RR, Weatherford T, Ross NM, Lamm RA, Menaker L. A modified gingival index for use in clinical trials. Clin Prev Dent. 1986 Jan-Feb;8(1):3-6. No abstract available. PMID 3485495